CLINICAL TRIAL: NCT05722912
Title: Expanded Access of Ruxolitinib Cream to Treat a Single Patient With cGVHD
Status: Approved for marketing | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I 18424-22-02
Record Dates: First submitted 2022-10-04; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: ruxolitinib; acute or chronic steroid-refractory GVHD; hematopoietic stem cell transplantation (allo-HSCT)
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib Cream
  Other Names: INCB018424

SUMMARY:
To provide ruxolitinib through an expanded access to treat a single patient with cGVHD

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Study Director — Children's Hospital Medical Center, Cincinnati